CLINICAL TRIAL: NCT01638741
Title: Rehabilitation and the Association With Attachment Styles Among Patients With Gynaecological Cancer
Brief Title: The Need for Rehabilitation and the Connection With Attachment Styles Among Patients With Gynaecological Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kamila Adellund Holt (Other)
Collaborators: University of Southern Denmark (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kamila Adellund Holt, Principal Investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: Rehabilitation
Record Dates: First submitted 2012-05-17; First posted 2012-07-12 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Needs for Rehabilitation; Adult Attachment Style; Quality of Life.; Depression; PTSD
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Rehabilitation goals of patients with gynaecological cancer. — Conversations with the nurse and supportive phone calls. Conversation are structured and placed 1 and 3 months after surgery. Phone calls are carried out at two and three months after surgery.

SUMMARY:
The purpose of this study is to provide new knowledge about:

* Integration of rehabilitation in a highly specialized gynaecological department.
* Development and testing of an individually adapted rehabilitation process.
* Needs for rehabilitation among women with gynaecological cancer.
* Connection between adult attachment style for women with gynaecological cancer and their quality of life, rehabilitation needs and symptoms of depression /PTSD.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of gynaecological cancer
* surgery for gynaecological cancer

Exclusion Criteria:

* do not speak Danish

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description * Patients referred to Odense University Hospital outpatient clinic with suspition for gynaecological cancer. The patients are from to Regions in Danmark, Region Zealand and Region South Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-06 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of life at 5 months after surgery. | at baseline and 5 months after surgery
  EORCT QLQ-C 30 (QLQ is quality of life questionnaire) and EORCT QLQ-OV28 (OV - Ovarian) and EORCT QLQ-EN ( EN - endometrial) 24 and EORCT QLQ- CX 24 ( CX - cervix.

SECONDARY OUTCOMES:
Change from baseline in Revised Adult Attachment at 5 months after surgery. | At baseline and 5 months after sugery
  Revised Adult Attachment Scale (RAAS- 18) is used to measure attachment style among women with gynaecological cancer.
Change from baseline in Depression at 5 months after surgery. | At baseline and 5 months after surgery.
  MDI-12 (Major Depression Inventory), ICD-10 (International Classification of Diseases), measure the depression level in the period from baseline and 5 months after surgery.
Change from baseline in Posttraumatic stress disorder at 5 months after surgery | At baseline and 5 months after surgery.
  To measure the Posttraumatic stress disorder we uge HTQ-17 (Harvard Trauma Questionnaire) for PTSD (Post Traumatic Stress Disorder).

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark